CLINICAL TRIAL: NCT00632463
Title: RI-001 in Immunosuppressed Respiratory Syncytial Virus (RSV) Infected Patients at Risk of Lower Tract RSV Illness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ADMA Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ADMA-001
Record Dates: First submitted 2008-03-03; First posted 2008-03-10 (Estimated); Results first posted 2013-04-24 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-03

CONDITIONS: Upper Respiratory Tract Infection; Lower Respiratory Tract Infection
Keywords: Transplant; Immunosuppression
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Dose regimen 1
  Interventions: Biological: RI-001
- 2 (Experimental): Dose regimen 2
  Interventions: Biological: RI-001
- 3 (Placebo Comparator): Placebo
  Interventions: Biological: RI-001

INTERVENTIONS:
Biological: RI-001 — Dose 1
  Arms: 1
Biological: RI-001 — Dose 2
  Arms: 2
Biological: RI-001 — Placebo
  Arms: 3

SUMMARY:
RSV infections can develop into serious, life threatening conditions among immunocompromised patients. The objective of this study (ADMA 001) is to evaluate the safety and efficacy of RI-001 for the prevention of lower respiratory tract infections in immunocompromised patients identified as being infected with RSV in the upper respiratory tract.

ELIGIBILITY:
Inclusion Criteria:

1. An IEC/IRB approved written informed consent signed and dated by the patient or by parent(s) or a legally acceptable representative. The consent form or a specific assent form, where required, will be signed and dated by minors.
2. Documented Bone Marrow Transplant (BMT)/Hematopoietic Stem Cell Transplant (HSCT), Pulmonary/Cardiac Transplant, Pulmonary Transplant or Liver Transplant within the 2 years prior to randomization to the study drug.
3. Male/Female patients age: (Pediatric) ≥2 years and <16 years at the time of informed consent.
4. Male/Female patients age: (Adult) ≥ 16 years and ≤ 65 years at the time of informed consent.
5. Patient must have an URTI as defined by Respiratory Assessment Score (RAS)=1.
6. Patients must be actively taking at least one immunosuppressive agent.
7. Patients must have a positive RSV RT-PCR at the time of the randomization procedures.
8. Female patients must be of non-childbearing potential or have a negative pregnancy test prior to study start and be deemed not at risk of becoming pregnant by adherence to a reliable contraceptive method for the duration of the study. Females of non-childbearing potential are defined as women who have had a hysterectomy, bilateral oophorectomy, tubal ligation or who have been post-menopausal for at least two years, or are considered to be sterile due to recent chemotherapy.
9. Female patients who are not breast-feeding.
10. Patient/legally acceptable representative considered as reliable and capable of adhering to the protocol (e.g. able to understand and complete diaries and questionnaires), visit schedules or treatment regimen according to the judgment of the Investigator.

Exclusion Criteria:

1. Documented RSV lower respiratory tract infection (respiratory assessment score is greater than 1) as determined by the site investigators or research staff.
2. Requirement for mechanical ventilation, extracorporeal membrane oxygenation, continuous positive airway pressure or other mechanical respiratory or cardiac support
3. Unstable respiratory status so severe that survival is not expected for longer than 6 months.
4. End organ dysfunction resulting in anticipated survival of less than 6 months.
5. Known to be HIV positive.
6. Administration of any RSV specific products, including palivizumab (Synagis®) in the 3 months prior to randomization procedures.
7. Previous, current, or planned administration of an investigational RSV vaccine.
8. Known hypersensitivity to immunoglobulin.
9. Known Immunoglobulin (IgA) deficiency
10. Known renal impairment requiring any form of dialysis (HD, PD, CRRT).
11. Known hemodynamically significant congenital heart disease.
12. Previous poor compliance with visit schedules.
13. Severe medical, neurological or psychiatric disorders or laboratory values which may have an impact on the safety of the patient.
14. Concurrent participation in other investigational drug product studies; any exception must be approved by the ADMA Biologics Medical Director.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Upton Allen, MBBS, Principal Investigator — Division of Infectious Diseases, Hospital for Sick Children, Toronto, Ontario, Canada
Locations (19):
- United States (15):
  - University of California San Francisco, San Francisco, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - All Children's Hospital, St. Petersburg, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - New England Medical Center, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Schneider Children's Hospital, New Hyde Park, New York
  - University of Rochester Medical Center, Rochester, New York
  - Oregon Health and Science University, Portland, Oregon
  - Children's Medical Center of Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Seattle Children's Hospital and Regional Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Canada (4):
  - Alberta Children's Hospital, Calgary, Alberta
  - Hospital for Sick Children, Toronto, Ontario
  - Hopital Maisonneuve Rosemont, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment period took place between 06Jun2008 and 05Mar2010. Patient recruitment took place in hospitals.
Groups:
- 1 (High Dose): Dose regimen 1 (High Dose): RI-001 1,500 mg/kg dose on day 1, and 750 mg/kg dose on day 3.
- 2 (Low Dose): Dose regimen 2 (Low Dose): RI-001 750 mg/kg dose on day 1, and 750 mg/kg dose on day 3.
- 3 (Placebo): Placebo (Normal saline): 7.5 mL/kg or 15 mL/kg dose on day 1, and 7.5 mL/kg dose on day 2.
Period: Overall Study
Arm/Group | 1 (High Dose) | 2 (Low Dose) | 3 (Placebo)
Started | 7 | 7 | 7
Completed | 7 | 6 | 7
Not Completed | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 (High Dose) | 2 (Low Dose) | 3 (Placebo) | Total
Number analyzed (Participants) | 7 | 7 | 7 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 2 | 2 | 7
  Between 18 and 65 years | 3 | 5 | 4 | 12
  >=65 years | 1 | 0 | 1 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 37 (29.06) | 33 (23.25) | 44.14 (25.06) | 38.04 (25.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 3 | 13
  Male | 2 | 2 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 7 | 4 | 6 | 17
  Canada | 0 | 2 | 0 | 2
  Australia | 0 | 1 | 0 | 1
  New Zealand | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Circulating RI-001 Titer
Description: The primary endpoint of this study was the mean fold titer increase from baseline to Day 18 in circulating serum anti-RSV neutralizing antibody following treatment with RI-001.
Time Frame: Study day 18
Measure: Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | 1 (High Dose) | 2 (Low Dose) | 3 (Placebo)
Number analyzed (Participants) | 7 | 7 | 7
Fold Change | 9.24 [4.07 to 21.02] | 4.85 [2.22 to 10.59] | 1.42 [0.64 to 3.17]

2. Secondary Outcome: Incidence of RSV Progression From Symptomatic Upper Respiratory Tract Infection to Lower Respiratory Tract Infection.
Time Frame: Study day 33
Measure: Number; unit: Participants
Arm/Group | 1 (High Dose) | 2 (Low Dose) | 3 (Placebo)
Number analyzed (Participants) | 7 | 7 | 7
Participants | 1 | 2 | 1

3. Secondary Outcome: The Number of Patients Achieving at Least a 4-fold Increase in Serum RSV Neutralizing Antibody Titers
Time Frame: 18 Days
Measure: Number; unit: Participants
Arm/Group | 1 (High Dose) | 2 (Low Dose) | 3 (Placebo)
Number analyzed (Participants) | 7 | 7 | 7
Participants | 6 | 3 | 0

ADVERSE EVENTS:
Arm/Group | 1 (High Dose) | 2 (Low Dose) | 3 (Placebo)
Serious Adverse Events (participants affected / at risk) | 2/7 | 4/7 | 1/7
Other Adverse Events (participants affected / at risk) | 4/7 | 6/7 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 (High Dose) (N=7) | 2 (Low Dose) (N=7) | 3 (Placebo) (N=7)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 (High Dose) (N=7) | 2 (Low Dose) (N=7) | 3 (Placebo) (N=7)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (4)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Dysguesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Labile blood pressure (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Graft versus host disease (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Panic Attack (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Crepitations (General disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Breath sounds abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Unfortunately enrollment in this study was suspended early due to slow accrual rates.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other